CLINICAL TRIAL: NCT06564948
Title: Improving Mental Health Treatment for Individuals in Crisis Interacting with the Criminal Justice System
Brief Title: Treatment for Individuals Interacting with the Criminal Justice System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Michigan State University (Other); Mount Auburn Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NCHATS R34-4
Record Dates: First submitted 2024-07-02; First posted 2024-08-21 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-10

CONDITIONS: Suicide Risk; Psychiatric Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics; Social Justice; Methods

STUDY DESIGN:
Intervention Model Description: Preliminary effectiveness of FSJS+Navigator model on suicide severity and clinical outcomes using CAT-SS/MH, mental health, and mental health treatment/criminal legal outcomes will be assessed. Assessments occur at baseline, 1, 3, and 6 months, providing key statistics (distribution, correlation of outcome over time, missingness) needed to inform a fully-powered Hybrid II trial. Improvement in medically treated suicide attempts and CAT-SS indicators will be assessed over time using repeated measures ANOVA. This study is a non-experimental longitudinal design comparing treatment group (FSJS+Navigator) to 2 control groups (FSJS Only and Treatment As Usual). We will assess the following as moderators of intervention effects: sex, race/ethnicity, past suicide attempt, past behavioral health treatment, Area Deprivation index, mental health professional shortage area score, per capita incarceration, and other area-level social determinants of health variables using stratified and DDD models.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment as usual (TAU) (Experimental): This arm will consist of 2160 eligible individuals identified to have had criminal legal involvement in Cambridge Health Alliance catchment area cities other than Cambridge (Everett, Somerville, Malden, Medford, Chelsea, Revere, Winthrop). Police departments in these Treatment as Usual cities have no programs that link police officers and clinicians to follow up on safety planning and services. These individuals will be identified as having police involvement between 2009 and 2019.
  Interventions: Other: Treatment as usual (TAU)
- Family and Social Justice Section (FSJS) (Experimental): Consists of 200 Cambridge Health Alliance Patients Ages 18-100 Individuals who have come into contact with the Cambridge Police Department (as identified in the Family and Social Justice Section data) between 2009 and 2019.
  Interventions: Other: Family and Social Justice
- FSJS + Navigator (Experimental): 40 patients recruited during the study period in the Cambridge Health Alliance Emergency Department (ED) Ages 18-100 Individuals who are brought into the ED under police supervision (excluding individuals currently incarcerated) involuntarily brought to the ED for psychiatric evaluation because they are considered to be a risk to themselves or others (MA Law 123(12)); or the subject of a police call for service for a mental health issue who are willingly admitted to the ED
  Interventions: Other: Family and Social Justice Service and Navigator (FSJS+Navigator) Intervention

INTERVENTIONS:
Other: Treatment as usual (TAU) — TAU patients will be identified using "targeted limited chart review methods" used in our prior studies, "scraping" clinical notes in the EHR for criminal justice involvement. Initial Identification terms, "police", "arrest", "court", "summons", "jail", and "crime" will be used to identify candidates for police involvement, downloading the sentence in which the keyword appeared and the sentence before and after. Next, an iterative process of editing of the search terms will be conducted to remove patients with negation of the keyword ("did not commit a crime"), and other sentence characteristics that generate false positives ("cardiac arrest"). Samples of the resulting dataset will be taken, accuracy assessed by examining the surrounding sentences, leading to further iterations and repetition of the process until a high level of accuracy is achieved.
  Arms: Treatment as usual (TAU)
Other: Family and Social Justice — Documentation and follow-up by the Cambridge Police Department (CPD) for all mental health-related police calls, including involuntary and voluntary Emergency Department admissions; Established partnerships with city departments, healthcare systems, clergy, courts, businesses, and mental health advocates to ensure timely engagement in mental health treatment and community-based services; Required 40 hours of officer crisis intervention training (CIT), and additional sessions on trauma- informed policing, mental health, procedural justice, race, and crisis negotiation; and Staffing of sworn and civilian staff including specially-trained officers designated to work with individuals living with mental illness, homelessness, and substance abuse.
  Arms: Family and Social Justice Section (FSJS)
Other: Family and Social Justice Service and Navigator (FSJS+Navigator) Intervention — The FSJS+Navigator intervention adds an Emergency Department (ED)-based Systems Navigator, a community health worker with lived experience (as family member or patient) with criminal justice and mental health systems, to the FSJS. This navigator will enhance communication between Cambridge Police Department (CPD), Cambridge Health Alliance (CHA), and community agencies by being the needed "point person" within the healthcare system (the FSJS intervention only has a CPD-based social worker) to maintain communication to improve mental health services and prevent deeper justice involvement. The Navigator engages with the FSJS process in step i) of the above sequence, engaging the patient in the CHA ED and obtaining consent. The Navigator then discusses the case with the presenting CPD officer, and relays critical information about the context of the service call to ED staff. Next, the Navigator will administer the baseline CAT-MH/SS and assess additional needs (employment, housing, food).
  Arms: FSJS + Navigator

SUMMARY:
The proposed Center will leverage burgeoning real-time data linkage capabilities among health systems, Medicaid payors, and criminal legal (e.g., jail booking data, jail release data) systems, to identify individuals coming in and out of jail for suicide assessment and prevention, and to better coordinate care across these disparate systems. This Center will advance the fields of suicide prevention and criminal legal system-based mental health by solving a well-known, central problem in both fields: the inability to track and intervene with individuals moving in and out of both and often multiple systems. The goal is near-term reductions in the U.S. suicide rate.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment as Usual (TAU) arm

   1. Cambridge Health Alliance (CHA) patients from the cities other than Cambridge considered to be in the "catchment area" of CHA (Everett, Chelsea, Somerville, Medford, Malden, and Winthrop)
   2. Ages 18-100
   3. Identified as having police involvement between 2009 and 2019. Treatment as Usual patients will be identified using "targeted limited chart review methods" used in our prior studies, "scraping" clinical notes in the Electronic Health Records for criminal justice involvement. Initial Identification terms, "police", "arrest", "court", "summons", "jail", and "crime" will be used to identify candidates for police involvement, downloading the sentence in which the keyword appeared and the sentence before and after. Next, an iterative process of editing of the search terms will be conducted to remove patients with negation of the keyword ("did not commit a crime"), and other sentence characteristics that generate false positives ("cardiac arrest"). Samples of the resulting dataset will be taken, accuracy assessed by examining the surrounding sentences, leading to further iterations and repetition of the process until a high level of accuracy is achieved.
2. Family and Social Justice Section (FSJS) arm

   1. Cambridge Health Alliance patients from Cambridge
   2. Ages 18-100
   3. Individuals who have come into contact with the Cambridge Police Department (as identified in the Family and Social Justice Section data) between 2009 and 2019.
3. Family and Social Justice Section plus Navigator (FSJS+Navigator) arm

   1. Recruited during the study period in the CHA ED
   2. Ages 18-100
   3. Individuals who are brought into the Emergency Department under police supervision (excluding individuals currently incarcerated)

      * involuntarily brought to the Emergency Department for psychiatric evaluation because they are considered to be a risk to themselves or others (MA Law 123(12)); or
      * the subject of a police call for service for a mental health issue who are willingly admitted to the Emergency Department

Exclusion Criteria

1. Treatment as Usual (TAU) arm

   1. Cambridge Health Alliance patients residing in the City Cambridge are excluded from the TAU arm
   2. Under the age of 18
   3. Individuals with no identified criminal legal system contact during the study time period (no criminal legal involvement found in the targeted limited chart review method).
   4. Any individual incarcerated at the Middlesex Jail/Prison that has not been released by the end of the period of data collection (December 31, 2019).
2. Family and Social Justice Section (FSJS) arm

   1. Cambridge Health Alliance patients outside of Cambridge will be excluded from the FSJS arm
   2. Under the age of 18
   3. Any individual incarcerated at the Middlesex Jail/Prison that has not been released by the end of the period of data collection (December 31, 2019)
3. Family and Social Justice Section plus Navigator (FSJS+Navigator) arm

   1. Under the age of 18
   2. Any individual who becomes incarcerated during the course of the study
   3. Individuals who enter the Emergency Department not under police supervision

      * For example, individuals will be excluded who voluntarily come to the ED seeking psychiatric care because they feel they may be a risk to themselves or others
      * Individuals brought to the ED from a jail or court ordered to the ED as an alternative to jail or prison

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Past-year medically treated suicide attempt at baseline and 12 months | Baseline and 12 months
  Number of participants with a past-year medically treated suicide attempt. This will be measured at baseline and 12 months will be collected using the electronic health record (EHR) data.
Suicide Severity and Behaviors using Computerized Adaptive Test Suicide Scale (CAT-SS) at Baseline and 12 Months | Baseline and 12 months
  The CAT-SS measures Severity of Suicide Risk will be assessed using CAT-SS, providing severity on a 0-100 point scale, and risk-stratification to negligible, intermediate and high risk. It is highly sensitive and specific to the Columbia Suicide Severity Rating Scale, and predicts future suicide events with high precision and accuracy.

SECONDARY OUTCOMES:
Number of Individual Interactions with the Criminal Legal System at Baseline and 12 Months | From enrollment through 12 months
  Number of calls about each individual to the Cambridge Police Department (CPD) Number of arrests Number of admissions to the Middlesex County Jail Repeat admission to the Middlesex County Jail
Number of Individual Interactions between Hospitals and the Criminal Justice System at Baseline and 12 Months | From enrollment through 12 months
  Number of involuntary hospitalizations that require Cambridge Police Department (CPD) interaction
Frequency of Healthcare Services Used by Patients at Baseline and 12 Months | From enrollment through 12 months
  Number of Emergency Department visits Number of behavioral health inpatient visits Number of behavioral health outpatient mental health (MH) visits

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No